CLINICAL TRIAL: NCT03617107
Title: Reverse Total Shoulder Arthroplasty: A Data Analysis on Patients Undergoing Reverse Total Shoulder Arthroplasty
Acronym: rTSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Orthopaedic Research & Innovation Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ORIF.004
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Osteo Arthritis Shoulders; Proximal Humeral Fracture; Rotator Cuff Tear; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Shoulder Fractures; Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: reverse total shoulder arthroplasty — reverse total shoulder arthroplasty

SUMMARY:
The purpose of this study is to evaluate reverse total shoulder arthroplasty patients preoperative objective measurements and operative objective measurements to determine if there is any effect to postoperative outcomes. Patients who were 18 years old or greater at the time of surgery were followed clinically and radiographically to determine best practice and optimal treatment and technique, risk and rate of complication, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. >18 years of age
3. Reverse TSA performed by principal investigator

Exclusion Criteria:

1. Non-English speaking
2. <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients of principal investigator receiving rTSA for any indication at St. Elizabeth Healthcare between January 1, 2010 and October 31, 2017 will be evaluated and included in the data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
total operative time | preoperative to up to 8 years postoperative
  minutes
amount of blood loss | preoperative to up to 8 years postoperative
  mls

SECONDARY OUTCOMES:
Patient Outcomes | preoperative to up to 8 years postoperative
  American Shoulder and Elbow Surgeon score to measure shoulder function and pain. Scale of 0-100, 100 being the best possible score
Patient Outcomes | preoperative to up to 8 years postoperative
  Simple Shoulder Test score to measure shoulder function. Scale from 0-12, 12 being the most functional.

CONTACTS AND LOCATIONS:
Overall Officials: R M Greiwe, MD, Principal Investigator — The Orthopaedic Research & Innovation Foundation
Locations (1):
- The Orthopaedic Research & Innovation Foundation, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided